CLINICAL TRIAL: NCT07099105
Title: Subcostal Single-port Versus Intercostal Multi-port Robotic Lobectomy for Non-small Cell Lung Cancer: A Single-centre Retrospective Propensity Matched Study
Brief Title: Subcostal Single-port Versus Intercostal Multi-port Robotic Lobectomy for Non-small Cell Lung Cancer
Acronym: SP vs MP robot
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, Professor, Korea University Guro Hospital
Other Study IDs: 2025GR0224
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SP group: Patients with non-small cell lung cancer who underwent single-port robotic lobectomy. All procedures were performed using the SP system via the subcostal approach.
- MP: Patients with non-small cell lung cancer who underwent multi-port robotic lobectomy. All procedures were performed using the Xi system via the intercostal approach.

SUMMARY:
The goal of this observational study is compared the perioperative outcomes of robotic lobectomy using the SP system via the subcostal approach with those of multi-port robotic lobectomy using the Xi system via the intercostal approach.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years who underwent RATS lobectomy for NSCLC at the Korea University Guro Hospital between January 2017 and December 2024

Exclusion Criteria:

* patients who underwent Viedo-assisted thoracic surgery lobectomy
* patients who underwent robotic lobectomy with other combined surgery
* patients who received neoadjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged > 18 years who underwent robotic lobectomy for non-small cell lung cancer at the Korea University Guro Hospital between January 2017 and December 2024. Patients were categorized into the SP and MP groups based on the surgical approach employed.
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperatively day 0,1,2,3
  Postoperative pain using visual analog scale (minimum =0, maximum=10), A lower value reflects a lesser degree of pain perception (lower scores mean a better outcome)

SECONDARY OUTCOMES:
chest tube duration | Perioperative
  Chest tube duration refers to the number of days a thoracic drain remains in situ following pulmonary surgery. The duration is measured in days (minimum: 1, maximum: no defined). Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Lee JH, Park TH, Kim HK. Robotic thoracic surgery using the single-port robotic system: Initial experience with more than 100 cases. J Thorac Cardiovasc Surg. 2024 Dec;168(6):1513-1522.e2. doi: 10.1016/j.jtcvs.2024.03.005. Epub 2024 Apr 28. PMID 38678475